CLINICAL TRIAL: NCT01000987
Title: Effect of Varenicline on Fixed-Dose Alcohol Administration in Participants With Alcohol Use Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Sherry McKee, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0907005525
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-01

CONDITIONS: Alcohol Reactivity
Keywords: alcohol; reactivity; smoking cessation medications
MeSH Terms: interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Experimental): varenicline 1mg/day or 2mg/day
  Interventions: Drug: varenicline
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — 1mg/day or 2 mg/day Subjects are at steady state medication levels. They are participating during the 4-week medication period of our ongoing study, NCT00580645.
  Other Names: Chantix
  Arms: varenicline
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is the examine the effect of varenicline on cognition to a high dose (0.08 g/dL) of alcohol (vs. placebo alcohol) over the ascending and descending limb of the blood alcohol curve.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older
* Able to read and write in English
* Smokers and nonsmokers
* Meet criteria for alcohol use disorders
* Currently enrolled in NCT00580645

Exclusion Criteria:

* Any significant current medical or psychiatric conditions that would contraindicate the consumption of alcohol
* Significant hepatocellular injury
* Positive test results at intake appointments on urine drug screens conducted for opiates, cocaine, or benzodiazepines
* Women who are pregnant or nursing
* Suicidal, homicidal, or evidence of severe mental illness
* Prescription of any psychotropic drug in the 30 days prior to study enrollment
* Blood donation within the past 8 weeks
* Individuals who are seeking treatment for drinking or smoking or who have attempted to quit drinking or smoking within the past 3 months
* Known allergy to varenicline or taking H2blockers
* Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current protocol
* Subjects likely to exhibit clinically significant alcohol withdrawal during the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, Yale Human Behavioral Pharmacology Laboratory, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the n=60 subjects who completed the parent study (NCT00580645), n=44 elected to also complete the current protocol.
Groups:
- 1 mg/Day Varenicline: varenicline 1mg/day
  varenicline: 1mg/day Subjects are at steady state medication levels. They are participating during the 4-week medication period of our ongoing study, NCT00580645.
- 2 mg/Day Varenicline: varenicline 2mg/day
  varenicline: 2mg/day Subjects are at steady state medication levels. They are participating during the 4-week medication period of our ongoing study, NCT00580645.
Period: Overall Study
Arm/Group | 1 mg/Day Varenicline | 2 mg/Day Varenicline | Placebo
Started | 12 | 15 | 17
Completed | 12 | 15 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 mg/Day Varenicline | 2 mg/Day Varenicline | Placebo | Total
Number analyzed (Participants) | 12 | 15 | 17 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (7.29) | 34.4 (12.6) | 35.3 (9.47) | 34.6 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 6 | 15
  Male | 7 | 11 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function as Measured by Omissions on the CPT
Description: Cognitive function was measured using the Continuous Performance Task (CPT). The CPT assess attention and response inhibition and the main outcome was number of omissions (the number of times the target was present, but the subject did not respond) errors in response to go and stop targets. Participants are presented with "stop" and "go" targets that appear on a computer screen. They are told to press the space bar (respond) to "go" targets and to avoid pressing the space bar when "stop" targets appear. Presented in the data table are the average number of omissions (the number of times the target was present, but the subject did not respond). Higher omission rates indicate a greater level of inattention (range 0-324).
Time Frame: Following 3 weeks of medication. The CPT task was performed at 60 minutes following alcohol or placebo beverage consumption.
Measure: Mean (Standard Error); unit: Number of Omissions
Arm/Group | 1 mg/Day Varenicline | 2 mg/Day Varenicline | Placebo
Number analyzed (Participants) | 12 | 15 | 17
Number of Omissions
  Alcohol | 1.78 (1.24) | 1.28 (1.11) | 4.76 (1.05)
  Control Beverage | 0.98 (1.24) | 0.62 (1.11) | 2.37 (1.05)

ADVERSE EVENTS:
Time Frame: During the 1-week medication titration period (Days 1-8) of the parent study (NCT00580645).
Description: All adverse events reported during 1 week medication period. Baseline reporting not controlled. Subjects were queried about the presence/absence of severity of common symptoms (>5% and twice the rate seen in placebo-treated subjects) associated with varenicline. Adverse events assessed on Days 1, 2, 5 and 8.
Arm/Group | 1 mg/Day Varenicline | 2 mg/Day Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 5/20 | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 mg/Day Varenicline (N=20) | 2 mg/Day Varenicline (N=20) | Placebo (N=20)
Constipation (Gastrointestinal disorders) | 1 | 2 | 0
Nausea/Vomiting (Gastrointestinal disorders) | 4 | 5 | 6
Dry Mouth (General disorders) | 2 | 2 | 7
Insomnia (General disorders) | 0 | 5 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1
Difficulty Breathing (General disorders) | 1 | 1 | 0
Shortness of Breath (General disorders) | 0 | 1 | 1
Tightness in Chest (Cardiac disorders) | 1 | 0 | 0
Abnormal Dreams (General disorders) | 1 | 3 | 2
Fast Heartbeat (Cardiac disorders) | 1 | 3 | 1
Suicidal Thoughts (General disorders) | 0 | 0 | 0
Erratic Behavior (General disorders) | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No